CLINICAL TRIAL: NCT02368028
Title: Oral Alkali Production and Caries Prevention in Children (Cross-sectional Component)
Status: Completed | Type: Observational
Sponsor: University of Florida (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Dental and Craniofacial Research (NIDCR) (NIH)
Responsible Party: Sponsor
Other Study IDs: 272-2012; K23DE023579 (NIH)
Record Dates: First submitted 2015-02-13; First posted 2015-02-20 (Estimated); Last update posted 2015-09-15 (Estimated); Status verified 2015-09

CONDITIONS: Dental Caries
Keywords: Plaque; Saliva; Dental Caries
MeSH Terms: conditions — Dental Caries; Plaque, Amyloid

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Saliva and Dental Plaque
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Caries Free: Participants who do not have caries (cavities) will have oral samples collected.
  Interventions: Other: Oral Samples
- Caries Active: Participants who do have caries (cavities) will have oral samples collected.
  Interventions: Other: Oral Samples

INTERVENTIONS:
Other: Oral Samples — Oral samples of saliva, dental plaque and DNA will be collected between the two groups.

SUMMARY:
The fact that dental caries remains a major public health problem mandates that oral-health researchers explore new strategies for assessment of caries risk, as well as for caries prevention and management. Dental caries occurs when acids produced by bacterial glycolysis of dietary carbohydrates causes demineralization of the tooth enamel. A major focus of caries research has been on identifying and characterizing acid-generating bacteria and the mechanisms of acid resistance. The purpose of this study is to investigate the type of bacteria that grows in the mouth and on teeth.

DETAILED DESCRIPTION:
This study will require only one visit. The study visit will last about one hour. At the study visit, parent-administered questionnaires will be used to collect information on the following: (a) the participant's demographic background (age, gender, and race), (b) socio-economic status (parents' income and housing condition), (c) participant's oral health practice (feeding histories, diet habits, oral hygiene measures, and dental attendance), and (d) systemic diseases. During the study visit, the participant's complete medical and dental history will be obtained and reviewed, and a dental exam will be performed in order to determine participants' caries status, and intraoral pictures may be taken of participants' teeth.

Participants will not be allowed to brush or clean teeth using any type of oral hygiene procedures for 8 hours prior to sample collection. Saliva and plaque (The solf white-yellowish material on the tooth surface) will be collected. The Investigator will use a small probe to measure the pH of the dental plaque that builds up on the teeth. The participant will be asked to dip one finger into a glass containing a buffer solution and the probe will be placed on the teeth from which plaque will be taken.

Dental plaque will be collected from the participants between the ages of 2 and 5 with at least two teeth and who allow the dental examination and the sample collection procedures to be done safely. Plaque samples will be collected by gently scrapping the tooth using a sterile instrument. If the participant does not have enough plaque samples, they will be asked to return on the following day. Saliva will be collected by using cotton swabs or by asking the participant to spit into a sterile plastic container.

ELIGIBILITY:
Inclusion Criteria:

* Age 2 to 5 years

Exclusion Criteria:

* Treated with antibiotics within the past 3 months
* taking any medication at the time of the study
* uses orthodontic appliance, and
* has performed oral hygiene procedures in the past 8 hour prior to the collection appointment.

Ages: 2 Years to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The study population will consist of unrelated children aged between 2 and 5 years with different levels of caries experience.
Sampling Method: Probability Sample
Enrollment: 131 (Actual)
Dates: Start 2015-03; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Arginolytic activity in oral samples | Day 1
  Oral samples, saliva and dental plaque, will be collected and their arginolytic activity wil be compared between the two groups.

SECONDARY OUTCOMES:
Type of oral bacteria | Day 1
  DNA and RNA samples will be extracted from saliva and dental plaque and the type of oral bacteria and their metabolism present on theses samples will be compared between the two groups.

OTHER OUTCOMES:
Oral health | Day 1
  Oral exam will be performed to determine the oral health or disease status of the participants.

CONTACTS AND LOCATIONS:
Overall Officials: Marcelle Nascimento, DDS, PhD, Principal Investigator — University of Florida
Locations (1):
- Dental Clinical Research Unit, University of Florida, Gainesville, Florida, United States

REFERENCES:
- [Result] Nascimento MM, Liu Y, Kalra R, Perry S, Adewumi A, Xu X, Primosch RE, Burne RA. Oral arginine metabolism may decrease the risk for dental caries in children. J Dent Res. 2013 Jul;92(7):604-8. doi: 10.1177/0022034513487907. Epub 2013 May 2. PMID 23640952